CLINICAL TRIAL: NCT01363531
Title: Clinical Trial for the Assessment of Delayed Antibiotic Treatment Strategies in the Non-complicated Acute Respiratory Tract Infections in General Practice
Brief Title: Clinical Trial for the Assessment of Delayed Antibiotic Treatment Strategies
Acronym: PDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDA study
Record Dates: First submitted 2011-05-18; First posted 2011-06-01 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-03

CONDITIONS: Pharyngitis; Acute Tonsillitis; Rhinosinusitis; Acute Bronchitis; Chronic Obstructive Pulmonary Disease
Keywords: Prescription; Antibiotic; Acute respiratory infections; Satisfaction; Perception; Pharyngitis and/or acute tonsillitis; Rhinosinusitis; Acute bronchitis; Acute exacerbation of chronic obstructive pulmonary disease (mild to moderate)
MeSH Terms: conditions — Pharyngitis; Rhinosinusitis; Bronchitis; Pulmonary Disease, Chronic Obstructive; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Direct antibiotic treatment (Active Comparator): The doctor gives to patient an antibiotic prescription for his respiratory infection, which he should start immediately.
  Interventions: Other: Antibiotic prescription strategies
- No antibiotic treatment (No Intervention): The doctor doesn't give to patient an antibiotic prescription for his respiratory infection.
- Delayed antibiotic prescription 1 (Experimental): The doctor gives to patient an antibiotic prescription for his respiratory infection with the advice to use it if needed, in case of worsening of symptoms or not improving.
  Interventions: Other: Antibiotic prescription strategies
- Delayed antibiotic prescription 2 (Experimental): The doctor leaves the antibiotic prescription, for the respiratory infection of the patient, at the reception of the primary care center 3 days after the first medical visit. This prescription can be collected by patient if he needed, in case of worsening of symptoms or not improving.
  Interventions: Other: Antibiotic prescription strategies

INTERVENTIONS:
Other: Antibiotic prescription strategies — The patients enrolled will be randomized between four treatment strategies or arms. Patients randomized to delayed treatment arms or direct treatment, doctors can choose the antibiotic that they consider appropriate depending on such local resistance or practice.
  Arms: Delayed antibiotic prescription 1; Delayed antibiotic prescription 2; Direct antibiotic treatment

SUMMARY:
The general hypothesis is that delayed antibiotic treatment strategies present similar effectiveness, when compared with non-prescription of antibiotics or the prescription of antibiotics, in the non-complicated acute respiratory tract infections.

DETAILED DESCRIPTION:
The aim of the PDA study is to assess the efficacy and safety of different delayed antibiotic prescribing strategies, compared to direct antibiotic treatment and no antibiotic treatment, for the treatment of non-complicated acute respiratory infections, in terms of symptoms duration and severity. Moreover, antibiotic consumption, patient satisfaction, efficacy perception and number of medical visits will be also assessed for each therapeutic strategy.

The PDA is a multicentric study, parallel, randomised controlled trial to compare four antibiotic prescribing strategies in the non-complicated acute respiratory tract infections. The trial will include acute pharyngitis and/or acute tonsillitis, rhinosinusitis, acute bronchitis and acute exacerbation of chronic obstructive pulmonary disease with (mild to moderate) in adults. The expected number of patients to be included in this trial is 600. Therapeutic strategies include: direct antibiotic treatment, no antibiotic treatment, and two delayed antibiotic prescribing strategies (prescription given to patient with advice to use a course of antibiotics if needed in case of worsening of symptoms or not improving, and prescription left at the reception of the primary care center 3 days after the first medical visit). Follow-up period will be one month. The primary outcome will be symptom duration and severity. Other outcomes included will be use of antibiotics, patient satisfaction, perception of antibiotic efficacy, complications, and number of medical visits.

ELIGIBILITY:
General Inclusion Criteria:

In this study can be enrolled adult patients with non-complicated acute respiratory tract infections, including pharyngitis and/or tonsillitis, rhinosinusitis, acute bronchitis and exacerbations of chronic obstructive pulmonary disease mild to moderate. The doctors include patients with these infections if they have reasonable doubts if the patients should treat with antibiotics

General Exclusion Criteria:

* Patients have participated in the PDA previously.
* Patients are severely affected or patients has been felt severely affected for a week (all time)
* Patients with symptoms and signs suggestive of serious illness or severely affected and/or complications (particularly pneumonia, mastoiditis, peritonsillar abscess, peritonsillar cellulitis, intraorbital or intracranial complications).
* Patients at high risk of serious complications due to prior comorbidity. This includes significant heart disease, lung, kidney, liver or neuromuscular, immunosuppression, cystic fibrosis.
* If the patient is over 65 years with acute cough and two or more of the following criteria or more than 80 years with acute cough and one or more of the following criteria:
* Hospitalization in the previous year
* Diabetes Type I or II
* History of heart failure
* Current use of oral corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Duration and severity of symptoms. | 30 days
  Patients completed a diary of symptoms.

SECONDARY OUTCOMES:
Antibiotic consumption at 30 days. | 30 days
  Self-reported by the patients and checked at the Regional Pharmacy's Units.
Patient satisfaction | 30 days
  Likert scale
Patients' belief in the efficacy of antibiotics | 30 days
  Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Alonso Coello, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] de la Poza Abad M, Mas Dalmau G, Moreno Bakedano M, Gonzalez Gonzalez AI, Canellas Criado Y, Hernandez Anadon S, Rotaeche del Campo R, Toran Monserrat P, Negrete Palma A, Munoz Ortiz L, Borrell Thio E, Llor C, Little P, Alonso-Coello P; Delayed Antibiotic Prescription (DAP) Group. Prescription Strategies in Acute Uncomplicated Respiratory Infections: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jan;176(1):21-9. doi: 10.1001/jamainternmed.2015.7088. PMID 26719947
- [Derived] de la Poza Abad M, Mas Dalmau G, Moreno Bakedano M, Gonzalez Gonzalez AI, Canellas Criado Y, Hernandez Anadon S, Rotaeche del Campo R, Toran Monserrat P, Negrete Palma A, Pera G, Borrell Thio E, Llor C, Little P, Alonso Coello P; Delayed Antibiotic Prescription (DAP) Working Group. Rationale, design and organization of the delayed antibiotic prescription (DAP) trial: a randomized controlled trial of the efficacy and safety of delayed antibiotic prescribing strategies in the non-complicated acute respiratory tract infections in general practice. BMC Fam Pract. 2013 May 19;14:63. doi: 10.1186/1471-2296-14-63. PMID 23682979